CLINICAL TRIAL: NCT06894017
Title: Patient Preferences on Same-day Bilateral Intravitreal Dexamethasone Injections
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Miklos Schneider MD, PhD, Senior Consultant, Rigshospitalet, Denmark
Other Study IDs: p-2024-16883
Record Dates: First submitted 2025-03-17; First posted 2025-03-25 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Informed Consent; Preference, Patient
Keywords: Intravitreal; dexamethasone; injections; implant; questionnaire; patient preference; bilateral
MeSH Terms: conditions — Patient Preference | interventions — Calcium Dobesilate; Dexamethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Ozurdex (dexamethasone) — Intravitreal dexamethasone implant (Ozurdex) given according to the recommendations by the manufacturer.
  Other Names: Intravitreal dexamethasone implant

SUMMARY:
Intravitreal injections with dexamethasone implant (Ozurdex®) provide a reasonable and long-lasting treatment option in the cases of diabetic macular edema, as well as macular edema resulting from retinal vein occlusion and noninfectious posterior uveitis. During the course of these diseases, both eyes may be affected and may need therapy. The treatment burden associated with frequent medical visits associated with treatments in both eyes and follow-ups can be significant for patients and caregivers alike. Same-session bilateral ophthalmic procedures have proven safe and cost-effective, with patients consistently expressing a strong preference for this approach, particularly in the cases of cataract surgery and anti-VEGF injections when given the choice. The safety profile of same-day bilateral dexamethasone injections aligns with those of unilateral injections.

This patient preference study will focus on addressing the practical aspects of same-day bilateral dexamethasone injections from the patients' perspective and aims to explore the impact of personal and socio-economic variables, and the overall perspective of patients on choosing same-day bilateral dexamethasone injections. Understanding and mitigating the challenges patients face can lead to a more patient-friendly and resource-saving approach. Based on the outcomes of this study, considerations may be made to introduce bilateral injections at our department, potentially optimizing patient experience and clinical resources.

The aim of the study is to establish patient preferences regarding the administration of intravitreal dexamethasone implant injections in both eyes on the same day, in the same session and to identify key motivating and limiting factors from the patients' perspective.

ELIGIBILITY:
Inclusion criteria

* Having received at least one intravitreal dexamethasone implant in either eye
* >18 years of age
* Capacity to comprehend and answer questions in Danish language
* Signed informed consent

Exclusion criteria

• No intravitreal dexamethasone implant received within the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Capital Region of Denmark who are treated at Rigshospitalet.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Preference to bilateral injections | Through study completion, an average of 9 months
  Proportion of patients preferring and not preferring same-day bilateral dexamethasone implant injections

SECONDARY OUTCOMES:
Reasons | Through study completion, an average of 9 months
  For preferring or not preferring same-day bilateral injections from the patient's perspective
Differences in patient characteristics | Through study completion, an average of 9 months
  Between preference groups in: Age, Sex, Previous injection count, Indication for intravitreal treatment (medical diagnosis), Complications of previous treatments, Ocular comorbidity (e.g. glaucoma, cataract, previous retinal detachment etc.), Systemic comorbidity
Differences in socio-economic variables between preference groups | Through study completion, an average of 9 months
  As in: Need for caregivers, Means of transportation, Transport distance, Active vs retired, Highest education level

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Schneider, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Ophthalmology, Rigshospitalet, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bridges JFP, de Bekker-Grob EW, Hauber B, Heidenreich S, Janssen E, Bast A, Hanmer J, Danyliv A, Low E, Bouvy JC, Marshall DA. A Roadmap for Increasing the Usefulness and Impact of Patient-Preference Studies in Decision Making in Health: A Good Practices Report of an ISPOR Task Force. Value Health. 2023 Feb;26(2):153-162. doi: 10.1016/j.jval.2022.12.004. PMID 36754539
- [Background] Lin TC, Tseng PC, Hsu TK, Huang HW, Huang YM, Lo WJ, Chao CY, Chung YC. Same-Day Bilateral Intravitreal Dexamethasone Implants for the Treatment of Diabetic Macular Edema. Ophthalmologica. 2023;246(3-4):238-244. doi: 10.1159/000532056. Epub 2023 Aug 8. PMID 37552956
- [Background] Kapoor KG, Colchao JB. SAFETY OF CONSECUTIVE SAME-DAY BILATERAL INTRAVITREAL DEXAMETHASONE IMPLANT (OZURDEX). Retin Cases Brief Rep. 2020 Spring;14(2):200-202. doi: 10.1097/ICB.0000000000000653. PMID 29155696
- [Background] Dinh RH, Moushmoush O, Kolyvas P, Jacobsen BA, Mathai M, Sanghavi K, Levinson JD, Do BK. Describing Adverse Events Associated with Bilateral Same-Day Intravitreal Dexamethasone Implants. Ophthalmic Surg Lasers Imaging Retina. 2022 Nov;53(11):612-618. doi: 10.3928/23258160-20221018-04. Epub 2022 Nov 1. PMID 36378615
- [Background] Malcolm J, Leak C, Day AC, Baker H, Buchan JC. Immediate sequential bilateral cataract surgery: patient perceptions and preferences. Eye (Lond). 2023 May;37(7):1509-1514. doi: 10.1038/s41433-022-02171-7. Epub 2022 Jul 20. PMID 35859120
- [Background] Mahajan VB, Elkins KA, Russell SR, Boldt HC, Gehrs KM, Weingeist TA, Stone EM, Abramoff MD, Liu D, Folk JC. Bilateral intravitreal injection of antivascular endothelial growth factor therapy. Retina. 2011 Jan;31(1):31-5. doi: 10.1097/IAE.0b013e3181ed8c80. PMID 21187731
- [Background] Dickman MM, Spekreijse LS, Winkens B, Schouten JS, Simons RW, Dirksen CD, Nuijts RM. Immediate sequential bilateral surgery versus delayed sequential bilateral surgery for cataracts. Cochrane Database Syst Rev. 2022 Apr 25;4(4):CD013270. doi: 10.1002/14651858.CD013270.pub2. PMID 35467755
- [Background] Sav A, King MA, Whitty JA, Kendall E, McMillan SS, Kelly F, Hunter B, Wheeler AJ. Burden of treatment for chronic illness: a concept analysis and review of the literature. Health Expect. 2015 Jun;18(3):312-24. doi: 10.1111/hex.12046. Epub 2013 Jan 31. PMID 23363080
- [Background] European Medicines Agency. Ozurdex. Accessed 21/11/2023, https://www.ema.europa.eu/en/medicines/human/EPAR/ozurdex